CLINICAL TRIAL: NCT03820271
Title: Construction of New Predictive Mathematical Models of Mortality in Decompensated Cirrhotic Patients Who Are Candidates for Liver Transplantation
Brief Title: New Prognostic Predictive Models of Mortality of Decompensated Cirrhotic Patients Waiting for Liver Transplantation
Acronym: SUPERMELD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: K170914J
Record Dates: First submitted 2019-01-18; First posted 2019-01-29 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Decompensated Cirrhosis; Liver Transplantation
Keywords: Liver transplantation; Predictive prognostic models; Decompensated cirrhosis

STUDY DESIGN:
Intervention Model Description: The pre-inclusion visit will be between 1 week and at the latest 2 days before the inclusion visit. The duration of the inclusion period is 24 months. After inclusion, samples at D5, D10 and D14 (additional samples) for sequential analysis of CRP and ammonemia and simple clinical reassessment will be scheduled for the period of hospitalization or routine consultations. Subsequent scheduled visits will take place quarterly until the transplant. Comprehensive nutritional , frailty and CT assessment of sarcopenia (psoas) by abdominal CT without contrast injection will be performed at 6 months as part of the protocol. Additional visits will be scheduled as part of the usual patient follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SuperMELD (Other)
  Interventions: Other: SuperMELD

INTERVENTIONS:
Other: SuperMELD — The population of this arm will consist of patients newly enrolled in the National Liver Transplantation Waiting List for decompensated cirrhosis, whose liver function and MELD score are assessed at enrollment and then routinely reassessed at least quarterly during the waiting phase.
  Patients will be followed from their listing to transplantation or discharge or death.

SUMMARY:
The MELD score is a predictive model of cirrhosis mortality used in France since 2007 to prioritize access to liver transplantation for patients enrolled in the national waiting list. The predictive value of this score was recently revised downward with a C index of the order of 0.65-0.67 and 20% of the patients enrolled for decompensated cirrhosis have access to liver transplantation by a subjective system of "expert component" independent of the MELD because of this lack of precision. The use of the MELD score to individually define access to the transplant should so be reconsidered. Recently new predictive models of cirrhosis mortality better than MELD have been developed and new mortality predictors independent of MELD have been published.

The goal of this study is to design prognostic predictive models of mortality for decompensated cirrhotic patients enrolled on the national liver transplant waiting list including known (MELD, MELD Na) as more recent (CLIF-C AD, CLIF - CACLF) predictive models and new objective predictors studied in combination in order to optimize the system of allocation of hepatic allografts in France.

The expected benefits of this search are twofold:

* At the individual level: The possibility for patients at high risk of death but with intermediate MELD score to be transplanted.
* Public health plan:

  * Improving the equity of graft allocation system.
  * Decreased mortality in the waiting list by improving the fairness and efficiency of the graft allocation system, a major public health issue

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old) newly registered on national waiting list with main diagnosis "cirrhosis"
* Patients enrolled on the national waiting list under the "national liver score" allocation scheme whether an expert component is considered or not
* Patients (or trusted person or family member or close relation if the patient is unable to express consent) who have been informed and signed their informed consent
* Patients affiliated to a health insurance scheme

Exclusion Criteria:

* Patients enrolled with decompensated cirrhosis associated with hepatocellular carcinoma
* Patients on AVK (INR and therefore MELD and CLIF scores uninterpretable)
* Vulnerable population (person under guardianship or curatorship or deprived of liberty by a judicial decision)
* Pregnant and / or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
predictive value of the new multivariate prognostic models in patients listed for decompensated cirrhosis | Month 3.
  Predictive value of mortality and drop out in the waiting list

SECONDARY OUTCOMES:
Individual predictive value of each of the new candidate predictors | Month 3. Month 6, Month 9, Month 12Month 12
  CRP, copeptin, NT-pro BNP, vitamin D, leucocytes, PMN/lymphocytes ratio, urinary NGal, cystatin C, frailty index, sarcopenia (abdominal tomodensitometry to measure the surface of psoas), caloric intake, encephalopathy (ammonia level, stroop application), and transferrin.
Complications predicted by each of the independent predictors | Month 3 Month 6, Month 9, Month 12.Month 12
  infection, renal dysfunction, encephalopathy, bleeding, ACLF
Added predictive value for mortality and drop out of new multivariate prognostic models on MELD (model end stage for liver disease) | Months 3, Month 6, Month 9, Month 12.
Evaluation of the predictive value of the CLIF (Chronic LIver Failure)-C (cirhosis) AD (Decompensation) score in decompensated cirrhotics listed without organ failure | Months 3, Month 6, Month 9, Month 12.
  death and drop out

CONTACTS AND LOCATIONS:
Overall Officials: Candy Estevez, Study Chair — APHP DRCI; Laetitia Gregoire, Study Chair — APHP URC
Locations (1):
- Pr Duvoux, Créteil, France

IPD SHARING:
Plan to Share IPD: No